CLINICAL TRIAL: NCT01216956
Title: Metabolic Effects of an 8 Week Niaspan Treatment in Patients With Abdominal Obesity and Mixed Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Michel Krempf, Institut National de la Santé Et de la Recherche Médicale, France
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NIASPAN-C05-36
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Insulin Sensitivity; Lipoproteins Metabolism; Non Esterified Fatty Acid Kinetics; Lipid Profile
Keywords: extended release nicotinic acid; non esterified fatty acid (NEFA); insulin resistance; Cholesteryl ester transfer protein (CETP); High density lipoprotein cholesterol
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release nicotinic acid (Experimental)
  Interventions: Drug: Extended-release nicotinic acid versus placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Extended-release nicotinic acid versus placebo

INTERVENTIONS:
Drug: Extended-release nicotinic acid versus placebo — Voluntary men with mixed dyslipidemia and abdominal obesity will receive extended release nicotinic acid. The dose of niaspan will be up-titrated for 3 weeks starting at 500 mg/d in order to reach 2g/d at start of week 4 dose which will be continued until the end of week 8. After a wash-out period of 3 weeks, they will receive placebo for 8 weeks. According to their randomization arm, subjects will receive either in first place placebo followed by extended release nicotinic acid or the opposite.

SUMMARY:
Nicotinic acid (Niacin) has been used for many years for the treatment of dyslipidemia. Indeed Niacin decreases triglycerides (TG) and low density lipoprotein cholesterol (LDL-c) but more importantly increases high density lipoprotein cholesterol (HDL-c). Although the drug has been used for so long, its precise mechanism of action remains elusive. The aim of this study was to characterise the metabolic changes induced by 8 week treatment with Niacin in dyslipidemic, overweight patients. The importance of the inhibition of lipolysis on the overall lipid effects of niacin will be studied. In order to get a very comprehensive view of all metabolic activities of niacin, this study will investigate the potential effects of niacin on Glucose metabolism, lipid and lipoprotein turnover, quantitative changes in lipoproteins and key enzymes involved in lipid metabolism.

DETAILED DESCRIPTION:
24 patients will be included in a double blind placebo controlled cross-over 8 week study comparing placebo to Niaspan (a long release formulation of niacin). In order to prevent any drop out linked to the flushing side effect of niacin, patient will take aspirin (300mg) prior to treatment throughout the study duration. The study will include at start and end of each arm, a full lipoproteins quantification as well as a measure of enzymes involved in lipid metabolism. On day 42 and 56 of each period, after an administration of either placebo or 500mg of immediate release niacin respectively, changes in plasma free fatty acid levels will be measured for 8hours in order to assess potential loss of activity of niacin over time upon chronic treatment with niaspan. Half of the patient will have an exploration of their glucose metabolism using hyperinsulinic clamp technique, whereas in the other half a metabolic turnover study using stable isotopes will focus on their lipoproteins, triglycerides and cholesterol handling. These explorations will be done at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 94cm
* Triglyceride concentration between 150mg/dL and 400mg/dL
* HDL-c < 60mg/dL
* Body mass index: 27 to 35 kg/m²

Exclusion Criteria:

* cancer
* diabetes mellitus
* hepatic, renal or digestive disorder
* hypertension
* chronic medical treatment interfering on lipids parameters

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Evolution of non-esterified fatty acid and triglycerides concentrations over time | After 42 and 56 days of placebo or nicotinic acid treatment
  Twelve hours after ingestion of chronic treatment, measures of non esterified fatty acid and triglycerides concentrations were carried out during 480 minutes to assess acute and chronic treatment effect on lipolysis and on triglyceride concentration.
  To appreciate both acute and chronic effects, subjects received medicinal supplements in addition to their chronic treatment:
  * On day 42, 500 mg of placebo to assess chronic nicotinic acid effect versus placebo effect
  * On day 56, 500 mg of immediate-release nicotinic acid (INA) to assess acute versus chronic nicotinic acid effect.

SECONDARY OUTCOMES:
Insulin sensitivity after treatment | After 53 days of placebo or nicotinic acid treatment
  Euglycemic Hyperinsulinemic clamp with glucose tracer infusion
Lipoproteins metabolism | After 53 days of placebo or nicotinic acid treatment
  Stable Isotopic tracer infusion (d3-leucine, 13C-acétate, d5-glycerol)
Lipid profile | Before and after placebo or nicotinic acid treatment
  Measure of lipoproteins (VLDL, IDL, LDL, HDL) - characterization of lipoprotein's subfraction Measure of enzymatic activity of cholesteryl ester transfer protein (CETP), phospholipid transfer protein (PLTP) and lecithin cholesterol acyl transferase (LCAT)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Krempf, PhD, MD, Principal Investigator — Institut National de la Santé Et de la Recheche Médiacle
Locations (1):
- Centre de Recherche en Nutrition Humaine, Nantes, France

REFERENCES:
- [Derived] Blanchard V, Ramin-Mangata S, Billon-Crossouard S, Aguesse A, Durand M, Chemello K, Nativel B, Flet L, Chetiveaux M, Jacobi D, Bard JM, Ouguerram K, Lambert G, Krempf M, Croyal M. Kinetics of plasma apolipoprotein E isoforms by LC-MS/MS: a pilot study. J Lipid Res. 2018 May;59(5):892-900. doi: 10.1194/jlr.P083576. Epub 2018 Mar 14. PMID 29540575
- [Derived] Ferchaud-Roucher V, Croyal M, Moyon T, Zair Y, Krempf M, Ouguerram K. Plasma Lipidome Analysis by Liquid Chromatography-High Resolution Mass Spectrometry and Ion Mobility of Hypertriglyceridemic Patients on Extended-Release Nicotinic Acid: a Pilot Study. Cardiovasc Drugs Ther. 2017 Jun;31(3):269-279. doi: 10.1007/s10557-017-6737-y. PMID 28752209